CLINICAL TRIAL: NCT01684397
Title: A Phase I/II Trial of Pazopanib Alternating With Bevacizumab in Treatment-Naive Metastatic Clear Cell Renal Cell Carcinoma Patients
Brief Title: Pazopanib Hydrochloride and Bevacizumab in Treating Patients With Previously Untreated Metastatic Kidney Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 191711; NCI-2012-01247 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13-069; I 191711 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2012-08-24; First posted 2012-09-13 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Clear Cell Renal Cell Carcinoma; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Bevacizumab; Immunoglobulin G; Disulfides; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (pazopanib hydrochloride and bevacizumab) (Experimental): Patients receive pazopanib hydrochloride PO on days 1-28 and bevacizumab IV over 30-90 minutes on days 36 and 50. Courses repeat every 70 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Other: Laboratory Biomarker Analysis; Drug: Pazopanib Hydrochloride; Other: Pharmacological Study

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pazopanib Hydrochloride — Given PO
  Other Names: GW786034B; Votrient
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of pazopanib hydrochloride and bevacizumab and to see how well they work in treating patients with previously untreated kidney cancer that has spread to other places in the body (metastatic). Pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Pazopanib hydrochloride may also stop the growth of tumor cells by blocking blood flow to the tumor. Monoclonal antibodies, such as bevacizumab, can prevent tumor growth by blocking the ability of tumor cells to grow and spread. Giving pazopanib hydrochloride together with bevacizumab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* I. To determine the safe phase II dose of this novel regimen. (Phase I)
* II. To determine the median progression free survival (PFS) from this novel regimen. (Phase II)

SECONDARY OBJECTIVES:

* To evaluate the safety and toxicity of the proposed regimen. (Phase I)
* To evaluate the response rate. (Phase I)
* To evaluate the pharmacokinetics of pazopanib (pazopanib hydrochloride). (Phase I)

  * To evaluate the vascular endothelial growth factor (VEGF) levels and myeloid derived suppressor cell (MDSC) levels at various time points and correlate with response. (Phase I)
  * To evaluate the safety and toxicity of this new regimen. (Phase II)
  * To evaluate the VEGF levels, interleukin (IL)-8 levels and MDSC levels at various time points and correlate with outcome. (Phase II)
  * To evaluate the PFS rate at 12 months. (Phase II)
* To evaluate overall survival. (Phase II)

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

Patients receive pazopanib hydrochloride orally (PO) on days 1-28, and bevacizumab intravenously (IV) over 30-90 minutes on days 36 and 50. Courses repeat every 70 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and Phase II patients are followed up by telephone every 12 months

ELIGIBILITY:
Inclusion Criteria:

* Biopsy/pathology-proven clear cell renal cell carcinoma (CCRCC) with metastases
* Have an Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Hemoglobin >= 10 gm/dL
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Total bilirubin =< upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< ULN
* International normalization ratio (INR) and activated partial thromboplastin time (aPTT) < 1.2 x ULN
* Serum creatinine < 1.5 mg/dL or if serum creatinine > 1.5 mg/dL then calculate creatinine clearance (CrCL) > 30 mL/min
* Urine protein to creatinine ratio =< 1 (if urine protein creatinine ratio is > 1, then a 24-hour urine total protein must be assessed; subjects will be ineligible if the 24-hour urine protein is found to be > 1 gm)
* Normal cardiac ejection fraction (> 50%) by multi gated acquisition scan (MUGA) or echocardiogram
* Have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria present
* Ability to swallow and retain oral medication
* Subjects of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Subject or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Subjects with known brain metastases should be excluded from this clinical trial
* Prior VEGF targeted therapies for renal cell carcinoma (RCC) including adjuvant or neoadjuvant treatments; in phase 1 only, one prior therapy with high dose IL-2 or anti-programmed cell death (PD)-1 compound alone or in combination with cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) targeting drug is allowed on the trial
* Subjects diagnosed with another cancer in the past 3 years; excluding basal cell carcinoma or squamous cell carcinoma, of skin which were completely cured by resection
* Concurrent use of another anti-cancer drug including an investigational anti-cancer agent
* Major surgery within 28 days prior to treatment or major surgery planned during the next 6 months
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic or psychiatric illness/social situations that would limit compliance with study requirements
* History of any of the following cardio-vascular condition:

  * Myocardial infarction (MI)
  * Unstable angina
  * Coronary artery bypass grafting (CABG)-unless patient had a negative stress test within 6 months of screening
  * Coronary angioplasty or stenting
  * Symptomatic peripheral arterial disease (PAD)
  * History of symptomatic chronic congestive heart failure (CHF)
  * History of cerebrovascular accidents including transient ischemic attacks (TIA)
  * Corrected QT interval (QTc) > 480 msec
  * Uncontrolled hypertension (systolic blood pressure [BP] > 150 mm Hg or diastolic BP of > 90 mm Hg); if the screening BP is elevated, adjustments in anti-hypertensives are permitted and a re-screening will be permitted for BP assessment with three consecutive values obtained 2 minutes apart; the 3 values have to be below 150/90 mm Hg for eligibility and can only be obtained after 2 days of the last change in anti-hypertensive medication; use of clonidine is not permissible for adjusting the BP during this period
* History of deep vein thrombosis (DVT) or pulmonary embolism (PE) in the past 6 months
* Subjects should not have packed red blood cells (PRBC) or platelet transfusion within 14 days of the screening
* Evidence of active bleeding or bleeding disorder
* Subjects currently on anti-coagulation therapy are not eligible
* Unable to discontinue the use of prohibited medications
* Pregnant or nursing female subjects
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the subject an unsuitable candidate to receive study drug
* Received an investigational agent within 30 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-11-21 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Median PFS (Phase II) | Up to 30 days post-treatment
  Distributions of continuous variables will be summarized with commonly used statistics (mean, standard deviation, median, etc.), with sub-group associations tested using the Wilcoxon Rank Sum test.
Optimal phase II dose, defined as the largest dose level at which less than 2 out of the 6 patients experienced dose-limiting toxicity, graded according to Common Terminology Criteria for Adverse Events version 4.0 (Phase I) | Up to 140 days
  The frequency of toxicities will be tabulated for the dose estimated to be the maximum-tolerated dose.

SECONDARY OUTCOMES:
Incidence of grade 3 or higher toxicities, graded according to CTCAE version 4.0 | Up to 30 days post-treatment
  Categorical variables will be summarized in contingency tables, with associations of interest assessed using Fisher's exact test. The frequency of toxicities will be tabulated by grade across all dose levels and courses.
Overall survival (Phase II) | From the date of study enrollment to the date of death from any cause, assessed up to 30 days post-treatment
  Will be obtained using Kaplan-Meier and Proportional Hazards methods.
PFS rate at 12 months (Phase II) | At 12 months
  Distributions of continuous variables will be summarized with commonly used statistics (mean, standard deviation, median, etc.), with sub-group associations tested using the Wilcoxon Rank Sum test.
Response rate according to RECIST 1.1 (Phase I) | Up to 30 days post-treatment

OTHER OUTCOMES:
IL-8 levels | Up to 30 days post-treatment
  Distributions of continuous variables will be summarized with commonly used statistics (mean, standard deviation, median, etc.), with sub-group associations tested using the Wilcoxon Rank Sum test.
MDSC levels | Up to 30 days post-treatment
  Distributions of continuous variables will be summarized with commonly used statistics (mean, standard deviation, median, etc.), with sub-group associations tested using the Wilcoxon Rank Sum test.
Pazopanib exposure as measured by pharmacokinetics parameters | Course 1 on day 1 at pre-dose, 2 hours, and 4 hours post-dose; day 15 at pre-dose and 2 hours post-dose; and day 29
VEGF levels | Up to 30 days post-treatment
  Distributions of continuous variables will be summarized with commonly used statistics (mean, standard deviation, median, etc.), with sub-group associations tested using the Wilcoxon Rank Sum test.

CONTACTS AND LOCATIONS:
Overall Officials: Saby George, Principal Investigator — Roswell Park Cancer Institute
Locations (5):
- United States (5):
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Karamanos Cancer Institute, Detroit, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin